CLINICAL TRIAL: NCT04906694
Title: A Randomized, Placebo-controlled Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Intranasal STI-2099 (COVI-DROPS™) in Outpatient Adults With COVID-19
Brief Title: Study to Evaluate a Single Intranasal Dose of STI-2099 (COVI-DROPS™) in Outpatient Adults With COVID-19 (US)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRP-COV-201US
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Covid19
Keywords: covid-19
MeSH Terms: conditions — COVID-19 | interventions — STI-2020

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVI-DROPS (Experimental): 10, 20, or 40 mg of COVI-DROPS administered intranasally
  Interventions: Biological: COVI-DROPS
- Placebo (Placebo Comparator): 2 mL administered intranasally
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: COVI-DROPS — COVI-DROPS is a fully human monoclonal antibody which is a neutralizing antibody to SARS-CoV-2
  Other Names: STI-2099
  Arms: COVI-DROPS
Drug: Placebo — Diluent solution
  Arms: Placebo

SUMMARY:
This is a double-blind study designed to investigate the efficacy, safety and PK of a single dose of COVI-DROPS or matched placebo in outpatient adults who have tested positive for COVID-19 and are either asymptomatic or have mild symptoms.

DETAILED DESCRIPTION:
Subjects will be randomized 1:1:1:1 to receive a single dose of COVI-DROPS 10 mg, COVI-DROPS 20 mg, COVI-DROPS 40 mg, or placebo in a double-blind manner. Investigational product (COVI-DROPS or placebo) will be administered once on Study Day 1. Subjects will be followed to Day 60.

ELIGIBILITY:
Inclusion Criteria:

* Positive for COVID-19 with any approved RT-PCR or rapid antigen test within 7 days of planned treatment
* Either have no COVID-19 symptoms (asymptomatic) or mild symptoms
* Must be willing and able to comply with all planned study procedures and be available for all study visits and follow-up as required by this protocol
* Subject must have provided written informed consent which includes signing the institutional review board or independent ethics committee approved consent form prior to participating in any study related activity
* Willing to follow contraception guidelines

Exclusion Criteria:

* In the investigator's opinion, has moderate or severe symptoms or rapidly progressive symptoms which are likely to progress such that a hospitalization is imminent (within 24-48 hours)
* Any medical condition that, in the Investigator's opinion, could adversely impact safety or key objectives of the study, particularly any intranasal pathology or disease process.
* Has a documented infection other than COVID-19
* Pregnant or lactating women who are breast feeding or planning on either during the study
* Has participated or is participating in a clinical research study evaluating COVID-19 convalescent plasma, monoclonal antibodies (mAbs) against SARS-CoV-2, or intravenous immunoglobulin (IVIG) within 3 months or less than 5 half-lives of the investigational product (whichever is longer) prior to the screening visit
* Has a high risk of progressing to severe COVID-19 per CDC's risk stratification (See: https://www.cdc.gov/coronavirus/2019-ncov/need-extra-precautions/people-with-medical-conditions.html)
* Is an immunocompromised subject even if previously fully vaccinated against COVID-19 or recovered from a prior COVID-19 infection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have COVID-19-related visit or hospitalization | Baseline through Day 29
  Proportion of subjects who have COVID-19-related urgent medically-attended visit, emergency department assessment or hospitalization through D29 = COVID-19-related visits or hospitalization (CRVHD29)

SECONDARY OUTCOMES:
Proportion of subjects alive and free of hospitalization ˃ 24h duration for acute COVID-19 illness management through D29 | Baseline through Day 29
  Proportion of subjects alive and free of hospitalization ˃ 24h duration for acute COVID-19 illness management through D29
Viral load change from baseline to D8 | Baseline to Day 8
  Viral load change from baseline to D8 based on RT-PCR determined COVID-19 viral titers (Log-10 copies/mL)
Change in WHO Clinical Progression Scale score | Baseline to Day 8 and Day 29
  Change in WHO Clinical Progression score at D8 and D29 (score of 0-10, with lower score meaning better outcome)
Viral load change from baseline to D29 | Baseline to Day 29
  Viral load change from baseline to D29, based on reverse-transcriptase polymerase chain reaction (RT-PCR) determined COVID-19 viral titres (Log-10 copies/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (18):
- United States (18):
  - Future Innovative Treatments, LLC, Colorado Springs, Colorado
  - Clinical Neuroscience dba CNS Healthcare, Jacksonville, Florida
  - Med-Care Research, Miami, Florida
  - Clinical Neuroscience Solutions Healthcare, Orlando, Florida
  - Precision Research Center, Tampa, Florida
  - Clinical Site Partners, Inc, Winter Park, Florida
  - Randomize Now, Peachtree City, Georgia
  - Revival Research Institute, Dearborn, Michigan
  - Quality Clinical Research, Omaha, Nebraska
  - Remington Davis, Columbus, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - WR-ClinSearch, Chattanooga, Tennessee
  - Advanced Medical Trials, Georgetown, Texas
  - Precision Comprehensive Clinical Research Solutions, Grapevine, Texas
  - Centex Studies Inc. Houston, Houston, Texas
  - LinQ, Pearland, Texas
  - Epic Research, Red Oak, Texas
  - Infectious Diseases Associates of Central Virginia, Lynchburg, Virginia